CLINICAL TRIAL: NCT07020793
Title: Efficacy of Green Subthreshold Laser Therapy in the Treatment of Chronic Central Serous Chorioretinopathy
Brief Title: Green Subthreshold Laser Therapy for Chronic Central Serous Chorioretinopathy.
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, MD, PHD, Federico II University
Other Study IDs: 05809855 Federico II
Record Dates: First submitted 2025-06-03; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: the Presence of Subretinal Fluid (SRF)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: green subthreshold laser therapy — The intervention consists of green subthreshold laser therapy delivered using the Norlase µSec™ Technology, a novel microsecond-pulsed laser platform specifically designed for retinal treatments.

SUMMARY:
Chronic Central Serous Chorioretinopathy (CSCR) is a vision-threatening retinal disorder characterized by persistent subretinal fluid due to choroidal vascular hyperpermeability and retinal pigment epithelium (RPE) dysfunction. This study evaluates the efficacy and safety of green subthreshold laser therapy using Norlase µSec Technology as a novel, tissue-sparing approach for treating chronic CSCR. By targeting RPE repair without inducing visible retinal damage, this technique aims to resolve subretinal fluid, restore retinal architecture, and improve visual function. This is the first study to report clinical outcomes with this specific laser platform in chronic CSCR management.

ELIGIBILITY:
Inclusion Criteria:

Subretinal fluid for more than three months, confirmed by multimodal imaging, diagnosis of chronic CSC in at least one eye.

Exclusion Criteria:

any evidence of choroidal neovascularization on multimodal imaging, as well as a history of previous photodynamic therapy (PDT) or focal laser treatment for CSC, prior diagnosis of ocular hypertension, glaucoma, and optic nerve disorders, presence of active retinal conditions such as vitreomacular traction, epiretinal membrane, diabetic retinopathy, or retinal vein occlusion, lens opacities that could interfere with retinal imaging or compromise visual acuity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes adult patients diagnosed with chronic Central Serous Chorioretinopathy (CSCR), defined by the presence of subretinal fluid (SRF) persisting for more than 4 months, as confirmed by optical coherence tomography (OCT)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
change in central foveal thickness | 3 months
  to evaluate changen in Central foveal tickness (CFT), assessed on OCT images by manually placing calipers between the internal limiting membrane and the outer boundary of the retinal pigment epithelium, before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- university of Naples Federico II, Naples, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided